CLINICAL TRIAL: NCT00138125
Title: Phase II Randomized Trial of Faslodex and Herceptin, Alone and Combined, in the First - Line Treatment of Hormone Receptor-Positive, HER-2/Neu-Overexpressing Metastatic Breast Cancer
Brief Title: Fulvestrant and/or Trastuzumab as First-Line Therapy in Treating Postmenopausal Women With Stage IV Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to low accrual
Sponsor: Translational Oncology Research International (Other)
Collaborators: University of California, Los Angeles (Other); Genentech, Inc. (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000439421; UCLA-0502057-01 (Other: UCLA IRB); TORI-B-04 (Other: UCLA); 441350-RI-78322 (Other Grant/Funding Number: Genentech and AstraZeneca); NCT00203437 (obsolete NCT alias)
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): see intervention description for details
  Interventions: Drug: Faslodex; Biological: Herceptin

INTERVENTIONS:
Drug: Faslodex — Administered IM at 500 mg on day 1 of cycle 1, followed by 500 mg on day 15 of cycle 1, then 500 mg on day 1 of each cycle thereafter.
Biological: Herceptin — Given at 4 mg/kg IV on day 1 (cycle 1) then 2mg/kg IV weekly

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using fulvestrant may fight breast cancer by lowering the amount of estrogen the body makes. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether giving fulvestrant together with trastuzumab is more effective than giving fulvestrant or trastuzumab alone in treating breast cancer.

PURPOSE: This randomized phase II trial is studying how well fulvestrant and/or trastuzumab works as first-line therapy in treating postmenopausal women with stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall objective response rate in postmenopausal women with estrogen receptor (ER)- and/or progesterone receptor (PR)-positive, HER2/neu-overexpressing stage IV breast cancer treated with first-line therapy comprising fulvestrant and/or trastuzumab (Herceptin®).

Secondary

* Compare the duration of response in patients treated with these regimens.
* Compare overall survival of patients treated with these regimens.
* Compare the antitumor activity of these regimens, in terms of time to disease progression, in these patients.
* Compare the clinical benefit of these regimens in these patients.
* Determine the safety and toxicity of these regimens in these patients.
* Correlate HER2/neu expression and ER and/or PR expression with response in patients treated with these regimens.

OUTLINE: This is a randomized, controlled, open-label, multicenter study. Patients are stratified according to prior adjuvant endocrine therapy (yes vs no). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive fulvestrant intramuscularly on days 1 and 15 of course 1 and then on day 1 only in all subsequent courses.
* Arm II: Patients receive trastuzumab (Herceptin®) IV over 30-90 minutes on days 1, 8, 15, and 22.
* Arm III: Patients receive fulvestrant as in arm I in combination with trastuzumab as in arm II.

In all arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 8 weeks.

PROJECTED ACCRUAL: A total of 120 patients (40 per treatment arm) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Female patient, postmenopausal, defined as a woman fulfilling any one of the following criteria:

  * Age 60 years or older
  * Age 45 years or older with amenorrhea for > 12 months with an intact uterus
  * Follicle-stimulating hormone and estradiol levels within post-menopausal range
  * Having undergone a bilateral oophorectomy
* Histologically or cytologically proven adenocarcinoma of the breast
* Subjects must have archived rumor tissue available to compare the clinical response with tumor expression of biomarkers, such as HER-2, ER and PR; archived tissue will be used to confirm HER-2, ER and PR status, but results will not be used to determine subject eligibility for the study
* HER2-positive disease
* ER-positive and/or PR-positive disease
* ECOG performance status 0-2
* Life expectancy > 24 weeks
* Left ventricular ejection fraction > lower limit of normal
* No prior chemotherapy, endocrine therapy, Herceptin, or other biologic or investigational therapy for metastatic breast cancer
* No more than two prior endocrine agents in the adjuvant setting as single- or sequential-therapy is permitted, but no prior Faslodex therapy is permitted. A 1-month treatment-free period is required prior to receiving the first dose of trial treatments
* Prior adjuvant chemotherapy is permitted
* Prior adjuvant Herceptin permitted
* At least 1 month since prior surgery, radiotherapy, or endocrine therapy, with complete recovery from the effects of these interventions
* Patients must have ended any hormone replacement therapy at least 1 month prior to receiving the first dose of trial therapy
* Patients treated with bisphosphonates may enroll, with heir bone lesions only assessable for disease progression
* Patient is accessible and willing to comply with treatment and follow-up
* Patient is willing to provide written informed consent prior to the performance of any study-related procedures
* Required laboratory values:

  * Absolute neutrophil count > 1.5 x 10^9/L
  * Hemoglobin > 10g/dL
  * Platelet count > 100 x 10^9/L
  * Creatinine < 2.0 mg/dL
  * Total bilirubin < 1.5 x upper limit of normal
  * AST and ALT < 2.5 x ULN

Exclusion Criteria:

* Prior chemotherapy, hormonal therapy, Herceptin or other investigational therapy for metastatic breast cancer
* Prior treatment with Faslodex
* Concurrent therapy with any other non-protocol anti-cancer therapy
* Current or prior history of brain metastases
* History of any other malignancy within the past 5 years, with the exception of non-melanoma skin cancer or carcinoma-in-situ of the cervix
* Clinically significant cardiovascular disease, New York Heart Association Class II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
* Prior exposure of > 360 mg/m2 doxorubicin or liposomal doxorubicin, > 120 mg/m2 mitoxantrone, > 90 mg/m2 idarubicin, or > 720 mg/m2 epirubicin
* Active, uncontrolled infection requiring parenteral antimicrobials
* The presence of any other medical or psychiatric disorder that, in the opinion of the treating physician, would contraindicate the use of the drugs in this protocol or place the subject at undue risk for treatment complications
* Inability to comply with the study protocol or follow-up procedures
* Known hypersensitivity to any of the drugs used in this protocol or to active or inactive excipients of Faslodex
* History of bleeding diasthesis
* Long-term anticoagulant therapy other than anti-platelet therapy, such as with warfarin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-04; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Pietras, MD, PhD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Cancer Care Associates Medical Group, Inc, Redondo Beach, California
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period from June 2005 - August 2008 at academic medical clinics and community medical clinics.
Groups:
- Faslodex + Herceptin: Faslodex : Administered IM at 500 mg on day 1 of cycle 1, followed by 500 mg on day 15 of cycle 1, then 500 mg on day 1 of each cycle thereafter.
  Herceptin : Given at 4 mg/kg IV on day 1 (cycle 1) then 2mg/kg IV weekly
Period: Overall Study
Arm/Group | Faslodex + Herceptin
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Faslodex + Herceptin
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Of the two treated patients on this trial, the records show that one patient who received Herceptin only completed 3 cycles of therapy, while the second patient who received Herceptin in combination with Faslodex completed 9 cycles of therapy. The last survival data collected from October to November 2008 showed that these two participants were alive at that time.
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Faslodex + Herceptin
Number analyzed (Participants) | 2
participants | 2

2. Secondary Outcome: Overall Objective Response Rate
Description: Two patients were treated on a truncated trial. Not enough data was generated for any analysis.
Time Frame: 5 years
Population: Two patients were treated on a truncated trial. Not enough data was generated for any analysis.
Arm/Group | Arm I
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Tumor Progression
Description: Two patients were treated on a truncated trial. Not enough data was generated for any analysis.
Time Frame: 5 years
Population: Two patients were treated on a truncated trial. Not enough data was generated for any analysis.
Arm/Group | Faslodex + Herceptin
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Response
Description: Two patients were treated on a truncated trial. Not enough data was generated for any analysis.
Time Frame: 5 years
Population: Two patients were treated on a truncated trial. Not enough data was generated for any analysis.
Arm/Group | Arm I
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: Two patients were treated on a truncated trial. Not enough data was generated for any analysis.
Time Frame: 5 years
Population: Two patients were treated on a truncated trial. Not enough data was generated for any analysis.
Arm/Group | Faslodex + Herceptin
Number analyzed (Participants) | 0

6. Secondary Outcome: Clinical Benefit (CR + PR + SD > 6 Months)
Description: Two patients were treated on a truncated trial. Not enough data was generated for any analysis.
Time Frame: 5 years
Population: Two patients were treated on a truncated trial. Not enough data was generated for any analysis.
Arm/Group | Faslodex + Herceptin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events reported between June 2005 and August 2008.
Arm/Group | Faslodex + Herceptin
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faslodex + Herceptin (N=2)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Trial terminated due to slow patient accrual.Study closed with two subjects enrolled to treatment phase.Slow accrual was due to specific requirements of study population limiting enrollment and possibly due to availability of study drugs in clinic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less